CLINICAL TRIAL: NCT03335228
Title: Assessment of the Safety and Efficacy of Intralesional Platelet Rich Plasma in Reducing Scalp Symptoms and Promoting Hair Growth in Frontal Fibrosing Alopecia
Brief Title: Platelet Rich Plasma for Frontal Fibrosing Alopecia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DERM-2020-28608
Record Dates: First submitted 2017-07-27; First posted 2017-11-07 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Frontal Fibrosing Alopecia
Keywords: platelet rich plasma, frontal fibrosing alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Eclipse Easy Spin for PRP Treatment (Experimental): Assessing the safety and efficacy of platelet rich plasma for treating frontal fibrosing alopecia. This will be accomplished by the production of platelet rich plasma by the Eclipse Easy Spin centrifuge. Subjects will receive treatment once a month for 6 months. Platelet rich plasma will be administered via injections into the affected areas of the scalp.
  Interventions: Device: Eclipse Easy Spin for PRP

INTERVENTIONS:
Device: Eclipse Easy Spin for PRP — Autologous platelet rich plasma is prepared from subject's blood with the Eclipse Easy Spin centrifuge and injected into affected areas.

SUMMARY:
The primary objective of this study is to assess the efficacy and safety of platelet rich plasma in reducing scalp symptoms and promoting hair growth in patients diagnosed with frontal fibrosing alopecia. Platelet rich plasma is an autologous blood product, and platelet rich plasma will be administered intralesionally for this study. The platelet rich plasma used for this study will be prepared using the Eclipse Easy Spin centrifuge.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the efficacy and safety of platelet rich plasma in reducing scalp symptoms and promoting hair growth in patients diagnosed with frontal fibrosing alopecia. The secondary objective of this study is subject self-assessment through the Dermatology Quality Life Index (DQLI) and Hair-Growth Assessment (HGA) as well as investigator-assessment from baseline. Platelet rich plasma is an autologous blood product, and platelet rich plasma will be administered intralesionally for this study. The platelet rich plasma used for this study will be prepared using the Eclipse Easy Spin centrifuge. The duration of this study for participants is 8 months, including an initial screening visit, 6 monthly treatment visits, and a follow-up visit. Subjects eligible for this study are those diagnosed with frontal-fibrosing alopecia via biopsy and clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 18 and older
* Diagnosed by a board-certified dermatologist with frontal fibrosing alopecia
* Scalp biopsy consistent with frontal fibrosing alopecia diagnosis
* Willing to use Head and Shoulders shampoo for the scalp while in study
* Willing to abstain from over the counter and prescription hair/scalp products other than those supplied in the study
* Willing to abstain from the use of non-steroidal anti-inflammatory medications, aspirin, St, John's Wart, and high doses of Vitamin E supplementation for 4 weeks
* Subjects must be capable of giving informed consent
* Stated willingness to comply with all study procedures and be available for the duration of the study
* For women with reproductive potential, a willingness to use methods of contraception that will prevent the subject from becoming pregnant during the study. Adequate contraception methods include hormonal methods used for two or more menstrual cycles before screening (eg. oral contraceptive pills, contraceptive patch, or contraceptive vaginal ring), barrier methods (eg, contraceptive sponge, diaphragm in conjunction with contraceptive foam or jelly, or condom in conjunction with contraceptive foam or jelly), intrauterine methods (IUD), sterilization (eg, tubal ligation or a monogamous relationship with a vasectomized partner) and abstinence

Exclusion Criteria:

* Current immunosuppression
* Oral treatment of FFA within the last 3 months (such as hydroxycholroquine, doxycycline, minocycline, acitretin, mycophenolate mofetil, cyclosporine, prednisone, rituximab, and pioglitazone etc.)
* History of other scalp/hair disease
* Current chemotherapy or radiation
* Propensity for keloids or hypertrophic scarring
* Autoimmune disorders
* Hematologic disorder or bleeding disorder
* Platelet dysfunction
* Use of anticoagulation therapy
* Active malignancy
* Use of intralesional or topical corticosteroids in the last 6 weeks
* Scalp atrophy
* Pregnant and/or breastfeeding
* Allergy or intolerance to triamcinolone
* Severe allergies manifested by a history of anaphylaxis, or history or presence of multiple severe allergies
* Medical problems including HIV, connective tissue disorder, PCOS, or untreated thyroid disease
* Any psychiatric or medical condition that in the opinion of the investigator will interfere with patient's ability to participate in the trial
* Current use of tanning beds or any active tanning
* Planned upcoming pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Changes in the LPPAI score from baseline | Baseline to 3 years
  Changes in LPPAI (LICHEN PLANOPILARIS ACTIVITY INDEX) Scale of of 0-4 0= None 4=Severe
Changes in the hair growth from baseline to the completion of the study • Change in hair growth from baseline to study completion via investigator assessment of scalp photography | Baseline to 3 years
  Changes in hair growth from baseline to study completion using scalp photography hair growth in patients diagnosed with frontal fibrosing alopecia

SECONDARY OUTCOMES:
self-assessment using the Dermatology Quality Life Index | Baseline to 3 years
  Subject self-assessment using the Dermatology Quality Life Index (DQLI)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota Department of Dermatology; Ronda Farah, MD, Principal Investigator — University of Minnesota Department of Dermatology
Locations (1):
- University of Minnesota Department of Dermatology, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No